CLINICAL TRIAL: NCT01391546
Title: An Open-label, Randomised, Comparative, Multicentre Study of the Immunogenicity and Safety of ZOSTAVAX When Administered by Intramuscular Route or Subcutaneous Route to Subjects of 50 Years of Age and Older
Brief Title: Immunogenicity and Safety Study of ZOSTAVAX Administered by Intramuscular or Subcutaneous Route to Participants Aged From 50 Years Old (V211-045)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V211-045; ZTV03C (Other: MCMVaccBV (SPMSD) Protocol Number); V211-045 (Other: Merck Protocol Number); 2009-012458-19 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ZOSTAVAX intramuscular (IM) route (Experimental): Single dose of 0.65 mL via IM injection
  Interventions: Biological: ZOSTAVAX
- ZOSTAVAX subcutaneous (SC) route (Active Comparator): Single dose of 0.65 mL via SC injection
  Interventions: Biological: ZOSTAVAX

INTERVENTIONS:
Biological: ZOSTAVAX — 1 dose 0.65 mL
  Other Names: V211

SUMMARY:
PRIMARY OBJECTIVES

Two co-primary objectives are:

* To demonstrate that the immunogenicity of ZOSTAVAX administered by intramuscular route (IM) is non-inferior to ZOSTAVAX administered by subcutaneous route (SC)
* To demonstrate that ZOSTAVAX administered by IM route induces an acceptable fold-rise of varicella zoster virus (VZV) antibody titre from pre to 4-week post-vaccination

SECONDARY OBJECTIVES

Immunogenicity objectives

* To evaluate the immunogenicity as measured by VZV antibody titre at 4 weeks following ZOSTAVAX administered by IM or SC route
* To evaluate the immune response as measured by a second assay, the VZV Interferon gamma Enzyme-linked immunospot (ELISPOT) at 4 weeks following ZOSTAVAX administered by IM or SC route

Safety objective

- To describe the safety profile of ZOSTAVAX administered by IM or SC route

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >=50 years
* Varicella history-positive or residence for >30 years in a country with endemic VZV infection

Exclusion Criteria:

* Febrile illness
* History of hypersensitivity or anaphylactoid reaction to any of the vaccine components
* Prior herpes zoster episode clinically diagnosed or exposure to varicella or herpes zoster within the 4 weeks prior to vaccination
* Prior receipt of varicella or zoster vaccine
* Active untreated tuberculosis
* Thrombocytopenia, any other coagulation disorder contraindicating intramuscular injection
* Receipt of medication / vaccine that may interfere with study assessments
* Known or suspected immune dysfunction
* User of recreational / illicit drugs or subject with alcohol abuse or dependence within the last year
* Any condition that might interfere with the interpretation of the study,

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2012-10-15 (Actual); Study Completion 2012-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Diez-Domingo J, Weinke T, Garcia de Lomas J, Meyer CU, Bertrand I, Eymin C, Thomas S, Sadorge C. Comparison of intramuscular and subcutaneous administration of a herpes zoster live-attenuated vaccine in adults aged >/=50 years: a randomised non-inferiority clinical trial. Vaccine. 2015 Feb 4;33(6):789-95. doi: 10.1016/j.vaccine.2014.12.024. Epub 2014 Dec 30. PMID 25555381

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Started | 177 | 177
Vaccinated | 176 | 177
Completed | 176 | 177
Not Completed | 1 | 0
Not completed — History of Herpes Zoster (HZ) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route | Total
Number analyzed (Participants) | 177 | 177 | 354
Age, Customized [Number; unit: Participants]
  50-59 years of age | 81 | 82 | 163
  60-69 years of age | 56 | 55 | 111
  ≥70 years of age | 40 | 40 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 97 | 195
  Male | 79 | 80 | 159
Age at Vaccination [Mean (Standard Deviation); unit: Years of Age] — Age of all vaccinated participants at Day 0 (time of vaccination) Population: One enrolled participant in IM arm withdrew prior to vaccination
  Years of Age
    number analyzed (Participants) | 176 | 177 | 353
    (all) | 62.6 (8.3) | 62.6 (8.5) | 62.6 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titre (GMT) of Varicella Zoster Virus (VZV) Antibodies 4 Weeks Post-vaccination
Description: Blood samples taken at 4 weeks post vaccination to determine the geometric mean titre (GMT) of VZV antibodies via Glycoprotein Enzyme Linked Immunosorbent Assay (gpELISA).
Time Frame: 4 week post-vaccination
Population: All randomised participants who had received the study vaccine, had at least one valid immunogenicity evaluation for VZV antibody and had post-vaccination data available for endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Number analyzed (Participants) | 168 | 173
gpELISA units/mL | 395.3 [350.6 to 445.6] | 391.7 [348.9 to 439.7]
Statistical Analysis 1: Comparison: ZOSTAVAX Intramuscular (IM) Route vs ZOSTAVAX Subcutaneous (SC) Route; Test type: Non-Inferiority or Equivalence — Non-inferiority was achieved if the lower bound of the 2-sided 95% confidence interval (CI) for the GMT ratio was greater than 2/3; p < 0.001, longitudinal regression model; Model adjusted for pre-vaccination titres and age at vaccination in years; GMT Ratio = 1.05, 95% CI 2-sided [0.93 to 1.18] — GMT ratio = GMT IM route divided by GMT SC route

2. Primary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titre: IM Route
Description: Blood sample taken at predose (Day 0) and 4 weeks post vaccination to determine the geometric mean titre (GMT) of VZV antibodies via gpELISA. The GMFR was calculated as GMT Post-dose/GMT Pre-vaccination
Time Frame: Pre-vaccination (Day 0) and 4 week post-vaccination
Population: All randomised participants who had received the study vaccine via IM route, had at least one valid immunogenicity evaluation for VZV antibody and had post-vaccination data available for endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ZOSTAVAX Intramuscular (IM) Route
Number analyzed (Participants) | 168
Ratio | 2.7 [2.4 to 3.0]
Statistical Analysis 1: Comparison: ZOSTAVAX Intramuscular (IM) Route; Acceptability was demonstrated if the lower bound of the two-sided 95% CI was >1.4; Test type: Superiority or Other; GMFR = 2.7, 95% CI 2-sided [2.4 to 3.0] — GMFR = GMT Post-vaccination/GMT Pre-vaccination

3. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titre: SC Route
Description: Blood sample taken at predose (Day 0) and 4 weeks post vaccination to determine the geometric mean titre (GMT) of VZV antibodies via gpELISA. The GMFR was calculated as GMT Post-vaccination/GMT Pre-vaccination
Time Frame: Pre-vaccination (Day 0) and 4 week post-vaccination
Population: All randomised participants who had received the study vaccine via SC route, had at least one valid immunogenicity evaluation for VZV antibody and had post-vaccination data available for endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ZOSTAVAX Subcutaneous (SC) Route
Number analyzed (Participants) | 172
Ratio | 2.5 [2.2 to 2.8]

4. Secondary Outcome: Geometric Mean Count (GMCs) of VZV Interferon Gamma ((IFN-γ) Enzyme-Linked ImmunoSpot (ELISPOT) Antibodies
Description: Blood samples taken 4 weeks post-vaccination to determine the IFN-γ ELISPOT GMC's. Results were reported as ELISPOT count/10^6 Peripheral Blood Mononuclear Cells (PBMC)
Time Frame: 4 week post-vaccination
Population: All randomised participants in the ELISPOT subset (predetermined protocol-defined sites) who had received the study vaccine and had valid post-vaccination data for endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISPOT count/10^6 PBMC
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Number analyzed (Participants) | 103 | 105
ELISPOT count/10^6 PBMC | 209.8 [175.2 to 251.3] | 195.7 [161.9 to 236.6]

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of IFN-γ ELISPOT Antibodies
Description: Blood samples taken pre-vaccination and 4 weeks post-vaccination to determine the IFN-γ ELISPOT GMFR.
Time Frame: Pre-vaccination (Day 0) and 4 week post-vaccination
Population: All randomised participants in the ELISPOT subset (predetermined protocol-defined sites) who had received the study vaccine and had valid pre- and post-vaccination data for endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Number analyzed (Participants) | 93 | 90
Ratio | 3.3 [2.8 to 3.9] | 3.4 [2.7 to 4.3]

6. Secondary Outcome: Percentage of Participants Who Report at Least 1 Injection-site Adverse Reaction
Description: Participants entered data into daily diary card regarding previously identified possible injection site reactions of erythema, injection site swelling or injection site pain for 1st 4 days post-vaccination. Additionally, injection site reactions not prompted on diary card (unsolicited) were collected up 28 days post-vaccination. All injection site reactions (solicited or unsolicited) were recorded.
Time Frame: up to 28 days after vaccination
Population: All vaccinated participants who had follow-up safety data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Number analyzed (Participants) | 176 | 177
Percentage of Participants | 34.1 [27.1 to 41.6] | 64.4 [56.9 to 71.4]

7. Secondary Outcome: Percentage of Participants Who Report at Least 1 Systemic Adverse Event
Description: An adverse event (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Adverse events that were considered systemic (not localized) were summarized. These events included rashes of interest: i.e. Varicella, Varicella-like rashes, Herpes zoster or shingles and Herpes zoster-like rashes and other systemic adverse events.
Time Frame: up to Day 28 after vaccination
Population: All vaccinated participants who had follow-up safety data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Number analyzed (Participants) | 176 | 177
Percentage of Participants | 23.3 [17.3 to 30.2] | 22.6 [16.7 to 29.5]

8. Secondary Outcome: Percentage of Participants Who Report at Least 1 Serious Adverse Event
Description: A serious adverse event (SAE) is any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgement. The percentage of participants who reported an SAE within 35 days of vaccination were recorded.
Time Frame: up to 35 days after vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Number analyzed (Participants) | 176 | 177
Percentage of Participants | 0.6 [NA to 3.1] | 1.1

ADVERSE EVENTS:
Time Frame: up to 35 days
Description: Safety population included all participants who received vaccine and had safety follow-up data available.
Arm/Group | ZOSTAVAX Intramuscular (IM) Route | ZOSTAVAX Subcutaneous (SC) Route
Serious Adverse Events (participants affected / at risk) | 1/176 | 2/177
Other Adverse Events (participants affected / at risk) | 59/176 | 112/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZOSTAVAX Intramuscular (IM) Route (N=176) | ZOSTAVAX Subcutaneous (SC) Route (N=177)
Hernia obstructive (General disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZOSTAVAX Intramuscular (IM) Route (N=176) | ZOSTAVAX Subcutaneous (SC) Route (N=177)
Injection site erythema (General disorders) | 29 (29) | 94 (94)
Injection site pain (General disorders) | 46 (46) | 70 (70)
Injection site pruritus (General disorders) | 3 (3) | 11 (11)
Injection site swelling (General disorders) | 24 (24) | 67 (67)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must first obtain written consent from Sponsor. If consent is given, all abstracts manuscripts, texts, or presentation, etc. will be sent to Sponsor for review and approval prior to their publication or presentation. Sponsor shall have sixty days to review these documents and may refuse to give its consent in part or whole for confidential reasons (including but not limited to intellectual property rights, whether patentable or not).